CLINICAL TRIAL: NCT02688920
Title: A Single-center, Observational, Intraluminal Imaging Study of Duodenal Layer Morphometry in Patients With and Without Type 2 Diabetes Undergoing Endoscopy of the Upper Gastrointestinal Tract
Brief Title: Intraluminal Imaging of Duodenal Layer Morphometry in Patients With and Without Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Victoria Gomez (Other)
Responsible Party: Sponsor-Investigator, Victoria Gomez, Gastroenterologist, Mayo Clinic
Organization: Mayo Clinic (Other)
Other Study IDs: 15-007742
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- With T2DM: Subjects with type 2 diabetes.
  Interventions: Procedure: EUS and OCT imaging
- Without T2DM: Subjects without type 2 diabetes
  Interventions: Procedure: EUS and OCT imaging

INTERVENTIONS:
Procedure: EUS and OCT imaging — Intraluminal imaging using endoscopic ultrasound and endoscopic optical coherence tomography

SUMMARY:
This observational study is conducted to determine how the duodenal layer thicknesses (mucosa, submucosa, and muscularis) vary with several factors in patients with and without type 2 diabetes.

DETAILED DESCRIPTION:
Study Objectives

1. To assess duodenal layer (mucosa, submucosa and muscularis) thickness differences between patients with and without type 2 diabetes using endoscopic ultrasound (EUS) and optical coherence tomography (OCT).
2. To assess duodenal layer thickness differences between patients with type 2 diabetes.
3. To assess duodenal layer thickness differences as a function of measurement location along the length of the duodenum.
4. To compare measurements obtained by endoscopic ultrasound, to those obtained by optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria:

* Patient is already scheduled for upper endoscopy with ultrasound or OCT, such as those with Barrett's esophagus.
* Patient is willing to sign an informed consent form.

Exclusion Criteria:

* Patient is not a candidate for endoscopy, EUS, or OCT, such as those with strictures, inflammatory disease or previous anastomosis of the esophagus or duodenum.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing previously scheduled routine endoscopy of the upper gastrointestinal tract.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2016-03; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Thickness of the duodenal mucosa using OCT, and EUS if possible | During imaging

SECONDARY OUTCOMES:
Thickness of the duodenal submucosa using OCT if possible, and EUS | During imaging

OTHER OUTCOMES:
Thickness of the duodenal muscularis using OCT if possible, and EUS | During imaging

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Gomez, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buchwald H, Estok R, Fahrbach K, Banel D, Jensen MD, Pories WJ, Bantle JP, Sledge I. Weight and type 2 diabetes after bariatric surgery: systematic review and meta-analysis. Am J Med. 2009 Mar;122(3):248-256.e5. doi: 10.1016/j.amjmed.2008.09.041. PMID 19272486
- [Background] Nagatake T, Fujita H, Minato N, Hamazaki Y. Enteroendocrine cells are specifically marked by cell surface expression of claudin-4 in mouse small intestine. PLoS One. 2014 Mar 6;9(6):e90638. doi: 10.1371/journal.pone.0090638. eCollection 2014. PMID 24603700
- [Background] Haboubi NY, Lee GS, Montgomery RD. Duodenal mucosal morphometry of elderly patients with small intestinal bacterial overgrowth: response to antibiotic treatment. Age Ageing. 1991 Jan;20(1):29-32. doi: 10.1093/ageing/20.1.29. PMID 2028847
- [Background] Maluenda C, Phillips AD, Briddon A, Walker-Smith JA. Quantitative analysis of small intestinal mucosa in cow's milk-sensitive enteropathy. J Pediatr Gastroenterol Nutr. 1984 Jun;3(3):349-56. doi: 10.1097/00005176-198406000-00008. PMID 6737178
- [Background] Rosch T, Lorenz R, Zenker K, von Wichert A, Dancygier H, Hofler H, Siewert JR, Classen M. Local staging and assessment of resectability in carcinoma of the esophagus, stomach, and duodenum by endoscopic ultrasonography. Gastrointest Endosc. 1992 Jul-Aug;38(4):460-7. doi: 10.1016/s0016-5107(92)70477-5. PMID 1511822
- [Background] Chang KJ, Katz KD, Durbin TE, Erickson RA, Butler JA, Lin F, Wuerker RB. Endoscopic ultrasound-guided fine-needle aspiration. Gastrointest Endosc. 1994 Nov-Dec;40(6):694-9. PMID 7859967
- [Background] Sivak MV Jr, Kobayashi K, Izatt JA, Rollins AM, Ung-Runyawee R, Chak A, Wong RC, Isenberg GA, Willis J. High-resolution endoscopic imaging of the GI tract using optical coherence tomography. Gastrointest Endosc. 2000 Apr;51(4 Pt 1):474-9. doi: 10.1016/s0016-5107(00)70450-0. PMID 10744825
- [Background] Gniuli D, Calcagno A, Dalla Libera L, Calvani R, Leccesi L, Caristo ME, Vettor R, Castagneto M, Ghirlanda G, Mingrone G. High-fat feeding stimulates endocrine, glucose-dependent insulinotropic polypeptide (GIP)-expressing cell hyperplasia in the duodenum of Wistar rats. Diabetologia. 2010 Oct;53(10):2233-40. doi: 10.1007/s00125-010-1830-9. Epub 2010 Jun 30. PMID 20585935